CLINICAL TRIAL: NCT02450929
Title: Prospective Clinical Evaluation of the Taperguard Endotracheal Tube
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Michael Aziz, Associate Professor, Oregon Health and Science University
Other Study IDs: Taperguard
Record Dates: First submitted 2015-05-14; First posted 2015-05-21 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Postoperative Pneumonia
Keywords: post operative; pneumonia; vascular; orthopedic; urologic; neurologic
MeSH Terms: conditions — Pneumonia; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Standard Barrel-Cuff ETT: Standard Barrel-Cuff ETT use in surgical patients
- Taperguard ETT: Taperguard ETT use in surgical patients

SUMMARY:
This protocol is designed to determine if a transition from barrel-shaped cuff designs to the Taperguard endotracheal tube (ETT) reduces the incidence of postoperative pneumonia in a prospective evaluation of a large general, vascular, orthopedic, urologic and neurologic surgical population. The protocol was originally developed as a quality assurance project to evaluate a practice change that took place December 1, 2012. Data regarding postoperative pneumonia and related factors will be reviewed for the 18 months prior to the practice change and compared to data from the 14.5 months following the change. Since the results may be of interest to a wider audience, we are converting the project to a research study that may be published in the future.

The study will include data from all adult patients who had surgery at OHSU between June 1, 2011 and February 15, 2014. We anticipate that we will enroll approximately 40,000 subjects (at least 22,000 in the pre-intervention group and at least 16,000 in the post-intervention group). Data will be gathered from the OHSU electronic medical record system (Centricity and Epic).

6. A multiple logistic regression analysis will be employed to determine the rates of pneumonia between the use of a standard barrel-cuff designed ETT and the Taperguard ETT for the defined group of surgical patients. The regression analysis would be adjusted for confounding variables including ASA status, age, use of paralytic, RSI with cricoid pressure, weight, pre-existing lung disease.

DETAILED DESCRIPTION:
Ventilator associated pneumonia (VAP) is a common complication from tracheal intubation and ventilation. The incidence of this complication is poorly defined but ranges to as high as 21% in surgical intensive care units.1-4 Efforts to reduce these events have evaluated various endotracheal tube (ETT) configurations and changes in clinical practice. Regarding endotracheal tubes, the use of supraglottic suctioning offers patient benefit.5-10 However, a definitive benefit for supraglottic suctioning exists only for patients with prolonged ventilation11. While there may be benefit to supraglottic suctioning for shorter periods of ventilation, the lower incidence of pneumonia in this group makes clinical evaluation less feasible.

The Taperguard tube™ (Covidien, Boulder, CO) is designed to prevent micro aspiration around channels that otherwise form with a barrel-shaped cuff. Laboratory evidence suggests less passage of fluid around the tube then conventional barrel-shaped cuffs (Batchelder, IARS Abstract 2010). Furthermore, a clinical model in pigs suggests less chemical injury from aspiration compared to a barrel shaped cuff (Lichtenthal, Abstract Critical Care 2010, 14(Suppl 1):P229). Human clinical studies are limited to data on reduced dye leakage compared to barrel-shaped cuffs (Mulier, ASA abstracts; D'Haese Acta Anaesthesiol Scand 2013).12

Currently, there is no evidence that patients with brief ventilation such as those undergoing routine surgery may benefit from actual outcomes with this tapered shape compared to regular tubes. Because the incidence of postoperative pneumonia in these patients is lower than those with prolonged ventilation, a large clinical data set would be necessary to evaluate any potential difference.

Since 2011, Oregon Health & Science University (OHSU) has been documenting patient clinical care in a comprehensive point-of-care electronic medical record system (Centricity, General Electric, Fairfield, CT; EPIC, Verona, WI). This information can be collated to provide easy access to co-morbidities, clinical interventions, and ICD-9 discharge codes. In addition, OHSU is part of the National Surgical Quality Improvement Project (NSQIP). OHSU has been a collaborator in this effort since 2006 and collects data on 1,400 patients annually for vascular and general surgery patients (IRB 4621).

The identified incidence of postoperative pneumonia in our NSQIP patients at OHSU is 1.9%. This incidence is slightly below the national NSQIP average and below the risk-adjusted expected rate of postoperative pneumonia. With a large surgical population and access to detailed quality data from our electronic medical record system, OHSU lends itself well to a clinical investigation to improve patient care. As investigators, we have extensive experience with management of data systems for detailing patient outcomes.13

On December 1, 2012, OHSU instituted a practice change to transition from endotracheal tubes with a barrel-shaped cuff design to the Taperguard tube for all surgical patients. A quality assurance program was set up to monitor patient outcomes, including postoperative pneumonia, before and after this practice change. The investigators have developed this protocol as an expansion of the quality assurance program, to determine how this practice change has affected patient outcomes.

This study is designed as a chart review to collect data from all adult surgical patients at OHSU for the 18 months prior to the practice change (June 1, 2011 - November 30, 2012) and compare it to data for all adult patients having surgery during the 14.5 months following the practice change (December 1, 2012 - February 15, 2014). Subjects will be excluded if anesthesia was provided using a Hi-Lo, double lumen, reinforced, or laser endotracheal tube or a laryngeal mask airway. Data will be collected from the OHSU electronic medical records (Centricity and EPIC). We will gather all ICD-9 discharge coding related to postoperative pneumonia and link it to pertinent information from the patient's anesthesia record, including demographic and surgical case information. Postoperative pneumonia will be defined using the NSQIP definition (listed at the end of this protocol).

We anticipate that we will enroll approximately 40,000 subjects in the study. The identified incidence of postoperative pneumonia at OHSU currently is 1.9%. A power analysis was conducted to determine a meaningful sample size in light of a predicted improvement in pneumonia outcomes. To demonstrate a risk reduction from 1.9% to 1.5% with 80% power and 0.05 significance, 22,000 patients would need to be enrolled in the pre-intervention group and 16,000 patients in the post-intervention group.

The primary source of data for this study is the electronic medical record. The NSQIP database may be used for comparison and verification of the data collected.

During the study period, there have been no active institutional changes to address postoperative pneumonia and none are anticipated in the near future. Anesthesia techniques are not undergoing any major changes to address pneumonia outcomes and compliance with prophylactic antibiotic administration is optimized at OHSU. Similarly, the intensive care units implement a "bundle" practice to reduce pneumonia that includes GI prophylaxis, tracheal suctioning, elevated head of bed positioning, sedation vacation with spontaneous breathing trial once a day, and targeted antibiotic therapy.

A multiple logistic regression analysis will be employed to determine the rates of pneumonia between the use of a standard barrel-cuff designed ETT and the Taperguard ETT for the defined group of surgical patients. The regression analysis would be adjusted for confounding variables including ASA status, age, use of paralytic, RSI with cricoid pressure, weight, pre-existing lung disease.

While patient benefit from potential reduced micro aspiration may be assumed from preliminary data, additional costs associated with this new technology are not warranted without evidence of patient care benefit or reduced patient care costs. The ultimate outcome desired when selecting endotracheal tube and ventilation strategy is a reduction in lung injury, morbidity, and reduced costs. Because this new technology offers potential benefit, it is imperative that a large-scale clinical study confirm the hypothesis that pneumonia is reduced by altering cuff design before a change in practice can be advocated. Estimates of cost-savings achieved from potential positive data can be constructed. In this manner, the Taperguard tube has potential to demonstrate savings for hospitals and improved patient care.

ELIGIBILITY:
Inclusion Criteria:

large general, vascular, orthopedic, urologic and neurologic surgical population

Exclusion Criteria:

n/a

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include data from all surgical patients enrolled in the National Surgical Quality Improvement Project (NSQIP) (IRB4621) who had surgery at OHSU between June 1, 2011 and May 31, 2014. We anticipate that we will enroll approximately 2500 subjects in each arm of the study.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2012-12-12 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
incidence of postoperative pneumonia in a large surgical population | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Aziz, MD, Principal Investigator — Oregon Health and Science University

REFERENCES:
- [Derived] Martini RP, Yanez ND, Treggiari MM, Tekkali P, Soelberg C, Aziz MF. Implementation of the TaperGuard endotracheal tube in an unselected surgical population to reduce postoperative pneumonia. BMC Anesthesiol. 2020 Aug 24;20(1):211. doi: 10.1186/s12871-020-01117-4. PMID 32838740